CLINICAL TRIAL: NCT07377370
Title: Patient-Related Factors Influencing Postoperative Pain After Gingival Graft Harvesting From the Palate: A Prospective Study
Brief Title: Factors Influencing Postoperative Pain After Gingival Graft Harvesting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2025-01
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; gingival graft; patient-related factors; palatal wound healing; psychological profile
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gingival graft harvesting from the palate (Other): Participants undergoing epithelial graft harvesting from the palate as part of mucogingival surgery. The palatal wound will be treated by placing collagen sponges and hemostatic sutures.
  Interventions: Procedure: Gingival graft harvesting from the palate

INTERVENTIONS:
Procedure: Gingival graft harvesting from the palate — An epithelial gingival graft will be harvested from the palate of patients requiring mucogingival surgery.

SUMMARY:
This prospective cohort study aims to evaluate patient-related, psychological, and clinical factors influencing postoperative pain following gingival graft harvesting from the palate. Consecutive adult patients requiring mucogingival surgery for root coverage or soft tissue augmentation around teeth or dental implants will be recruited at the Clínica Universitària d'Odontologia of Universitat Internacional de Catalunya (Barcelona, Spain).

All participants will undergo standardized pre-surgical periodontal care and oral hygiene instruction prior to surgery. Gingival grafts will be harvested from the palate under local anesthesia using a standardized surgical technique. Postoperative management will include analgesic medication, antiseptic rinses, and standardized postoperative instructions.

Patient-reported outcomes will be collected using validated questionnaires to assess anticipated pain, postoperative pain, stress, dental anxiety, psychological profile, personality traits, pain catastrophizing, coping strategies, oral health-related quality of life, and analgesic consumption. Postoperative pain and discomfort during eating will be recorded daily for two weeks. Clinical variables, including palatal thickness, graft dimensions, operative time, operator experience, and donor-site wound healing, will also be assessed.

The primary outcome is postoperative pain intensity following palatal graft harvesting. Secondary outcomes include operative time, donor-site discomfort, oral health-related quality of life, analgesic consumption, psychological and behavioral factors, and donor-site healing. The results of this study aim to improve understanding of factors associated with postoperative pain and to support individualized patient management in mucogingival surgery.

DETAILED DESCRIPTION:
This prospective cohort study is designed to investigate patient-related, psychological, and clinical factors influencing postoperative pain following gingival graft harvesting from the palate. The study will be conducted at the Clínica Universitària d'Odontologia of Universitat Internacional de Catalunya (UIC), Barcelona, Spain, in accordance with the Declaration of Helsinki (October 2024 revision). The study protocol and informed consent will be reviewed and approved by the Ethical Committee of Universitat Internacional de Catalunya.

Consecutive adult patients requiring mucogingival surgery for root coverage or soft tissue augmentation around teeth or dental implants will be screened for eligibility. Inclusion criteria include systemically healthy individuals aged 18 years or older, a healthy periodontal status according to the AAP/EFP definition, and full-mouth plaque and bleeding scores ≤20%. Exclusion criteria include pregnancy or lactation, smoking ≥10 cigarettes per day, systemic or metabolic diseases affecting wound healing, use of medications interfering with healing, chronic pain disorders, psychiatric diagnoses, regular use of analgesics or psychotropic medications, allergy to ibuprofen, recent grafting procedures, and ongoing orthodontic treatment.

Prior to surgery, all patients will complete initial periodontal therapy when indicated, followed by professional prophylaxis and individualized oral hygiene instruction at least two weeks before the surgical procedure. On the day of surgery, gingival graft harvesting will be performed under local anesthesia using 4% articaine with epinephrine (1:100,000). An epithelialized gingival graft will be harvested from the palate using a standardized technique. Graft dimensions will be determined based on clinical requirements. In cases of bilaminar techniques, the graft will be de-epithelialized extra-orally, whereas the epithelium will be preserved for free gingival graft procedures. Donor-site management will include placement of collagen sponges and hemostatic sutures using non-resorbable suspensory mattress sutures.

All surgical procedures will be performed by postgraduate students enrolled in the Master's Degree in Periodontology at UIC. Operator experience will be recorded based on the year of residency. Postoperative care will be standardized for all participants and will include instructions to avoid mechanical trauma at the surgical site, prescription of ibuprofen 600 mg three times daily for five days, chlorhexidine mouth rinses for two weeks, and rescue medication with paracetamol if needed. Sutures will be removed after two weeks.

Sociodemographic data will be collected during the pre-surgical visit, including age, sex, education level, occupation, smoking habits, alcohol consumption, and body mass index. Patient-reported outcomes will be assessed using validated questionnaires evaluating anticipated pain, stress levels, dental anxiety, psychological profile, personality traits, pain catastrophizing, coping strategies, and previous grafting experience. Postoperative pain intensity and discomfort during eating will be recorded daily for two weeks using visual analog scales. Oral health-related quality of life will be assessed at baseline, one week, and two weeks postoperatively using the OHIP-5 questionnaire. Analgesic consumption during the first postoperative week will also be recorded.

Clinical variables will include palatal thickness measured by transgingival probing, graft dimensions recorded at the time of harvesting, total operative time, and duration of donor-site preparation. Donor-site wound healing will be evaluated at one and two weeks postoperatively using standardized clinical photographs assessed independently by two blinded examiners. A modified wound healing score will be applied, and inter-rater reliability will be calculated.

The primary outcome of the study is postoperative pain intensity following palatal gingival graft harvesting. Secondary outcomes include operative time, donor-site discomfort, oral health-related quality of life, analgesic consumption, psychological and behavioral factors, palatal thickness, graft dimensions, operator experience, and donor-site wound healing. The findings of this study aim to identify factors associated with postoperative pain and to support improved patient-centered management strategies in mucogingival surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mucogingival surgery for gingival augmentation or root coverage purposes
* Systemically healthy individuals aged 18 years or older
* Healthy periodontal status according to the AAP/EFP definition
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) ≤ 20%

Exclusion Criteria:

* Pregnancy or lactation
* Self-reported smoking ≥10 cigarettes/day
* Presence of metabolic or systemic diseases that negatively affect soft tissue healing
* Use of medications that may interfere with wound healing
* Chronic pain disorders (e.g., fibromyalgia)
* Psychiatric diagnoses
* Regular use of analgesics, antidepressants, anxiolytics, or opioids
* Allergy to the study medication (Ibuprofen)
* History of grafting within the past 6 months
* Ongoing orthodontic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 14 days post-surgery, recorded daily
  Postoperative pain will be assessed as pain intensity measured using a Visual Analog Scale (VAS). The VAS consists of a 100-mm horizontal line, where 0 mm indicates no pain and 100 mm indicates worst imaginable pain. Pain will be self-reported by patients once daily during the 14-day postoperative period.
  Unit of Measure: Pain intensity (millimeters on a 0-100 mm Visual Analog Scale)

SECONDARY OUTCOMES:
Total operative time | At the time of surgery
  Total operative time will be measured as the duration of the surgical procedure from the first incision to the completion of the final suture. Time will be recorded in minutes using a standard surgical timer. Longer times indicate longer procedures.
  Unit of Measure: Minutes
Duration of donor site preparation | At the time of surgery
  Duration of donor site preparation will be measured as the time from the initial incision at the donor site to completion of tissue harvesting and hemostasis. Time will be recorded in minutes using a standard surgical timer. Longer times indicate longer donor site preparation.
  Unit of Measure: Minutes
Discomfort at eating | 14 days post-surgery, recorded daily
  Discomfort while eating will be assessed using a 100-mm Visual Analog Scale for Discomfort (VAS). Patients will mark a point on a 100-mm horizontal line, where 0 mm indicates no discomfort and 100 mm indicates worst imaginable discomfort. Higher scores indicate greater discomfort while eating. Discomfort will be self-reported once daily for 14 days following surgery.
  Unit of Measure: Millimeters (0-100) on the Visual Analog Scale for Discomfort
Oral Health Impact Profile - 5 items (OHIP5) | Baseline and 2-weeks post-surgery
  Oral health-related quality of life will be assessed using the Oral Health Impact Profile - 5 items (OHIP-5) questionnaire. The OHIP-5 consists of 5 items, each scored from 0 to 4, where 0 = never and 4 = very often, for a total score range of 0-20. Higher scores indicate worse oral health-related quality of life. The questionnaire will be completed preoperatively and at 14 days post-surgery.
  Unit of Measure: Points (0-20) on the OHIP-5 questionnaire
Analgesic consumption | During the first week
  Postoperative analgesic consumption will be measured as the number of standard doses of pain medication taken by the patient during the 7-day postoperative period. Patients will record each dose taken in a daily diary, including the type and amount of analgesic. Higher numbers indicate greater analgesic use.
  Unit of Measure: Number of doses (or tablets/capsules)
Anticipated pain | Baseline
  Anticipated postoperative pain will be assessed using the Visual Analog Scale for Pain (VAS). Patients will mark a point on a 100-mm horizontal line, where 0 mm indicates no expected pain and 100 mm indicates worst imaginable expected pain. Higher scores indicate greater anticipated pain. This assessment will be completed preoperatively, immediately before surgery.
  Unit of Measure: Millimeters (0-100) on the Visual Analog Scale for Pain
Stress level (PSS-4) | Baseline
  Perceived stress will be assessed using the Perceived Stress Scale - 4 item version (PSS-4). The PSS-4 consists of 4 items, each scored from 0 to 4, where 0 = never and 4 = very often, for a total score range of 0-16. Higher scores indicate higher perceived stress. The questionnaire will be completed preoperatively, immediately before surgery.
  Unit of Measure: Points (0-16) on the Perceived Stress Scale - 4 item version (PSS-4)
Dental Anxiety (IDAF-4C) | Baseline
  Dental anxiety will be assessed using the Index of Dental Anxiety and Fear - Core 4 items (IDAF-4C). The IDAF-4C consists of 4 items, each scored from 1 to 5, where 1 = no anxiety and 5 = extreme anxiety, for a mean score range of 1-5. Higher scores indicate greater dental anxiety. The questionnaire will be completed preoperatively, immediately before surgery.
  Unit of Measure: Mean score (1-5) on the Index of Dental Anxiety and Fear - Core 4 items (IDAF-4C)
Psychological profile (SCL-90-R) | Baseline
  Psychological symptoms will be assessed using the Symptom Checklist - 90 Revised (SCL-90-R). The SCL-90-R consists of 90 items, each scored from 0 to 4, where 0 = not at all and 4 = extremely, for a Global Severity Index (GSI) score range of 0-4. Higher scores indicate greater psychological symptom severity. The questionnaire will be completed preoperatively, immediately before surgery.
  Unit of Measure: Mean score (0-4) on the Global Severity Index of the Symptom Checklist - 90 Revised (SCL-90-R)
Personality traits (BFI-10) | Baseline
  Personality traits will be assessed using the Big Five Inventory - 10 items (BFI-10). The BFI-10 consists of 10 items, each scored from 1 to 5, where 1 = disagree strongly and 5 = agree strongly, for a mean score range of 1-5 on each of the five personality domains (Extraversion, Agreeableness, Conscientiousness, Neuroticism, Openness). Higher scores indicate stronger expression of the respective personality trait. The questionnaire will be completed preoperatively, immediately before surgery.
  Unit of Measure: Mean score (1-5) for each domain on the Big Five Inventory - 10 items (BFI-10)
Pain Catastrophizing Scale (PCS) | Baseline
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS). The PCS consists of 13 items, each scored from 0 to 4, where 0 = not at all and 4 = all the time, for a total score range of 0-52. Higher scores indicate greater levels of pain catastrophizing. The questionnaire will be completed preoperatively, immediately before surgery.
  Unit of Measure: Total score (0-52) on the Pain Catastrophizing Scale (PCS)
Coping strategies (Brief COPE) | Baseline
  Coping strategies will be assessed using the Brief COPE questionnaire. The Brief COPE consists of 28 items across 14 subscales, each scored from 1 to 4, where 1 = I haven't been doing this at all and 4 = I've been doing this a lot. Higher scores indicate greater use of the respective coping strategy. The questionnaire will be completed preoperatively, immediately before surgery.
  Unit of Measure: Score (1-4) for each subscale on the Brief COPE questionnaire
Past grafting experience | Baseline
  Past grafting experience will be assessed by asking patients whether they have previously undergone gingival or soft tissue grafting procedures. Responses will be recorded as Yes or No.
  Unit of Measure: Categorical (Yes/No)
Palatal thickness | Baseline
  Palatal thickness will be measured at the donor site using an endodontic spreader with a stop. The measurement will be recorded in millimeters (mm) at the level of the premolars on the hard palate. Higher values indicate a thicker palatal tissue.
  Unit of Measure: Millimeters (mm)
Graft dimensions | At the time of surgery
  Graft dimensions will be measured immediately after harvesting. Length, width, and thickness of the graft will be recorded in millimeters (mm) using a periodontal probe (PCP15). Higher values indicate larger graft size.
  Unit of Measure: Millimeters (mm) for length, width, and thickness
Operator experience | At the time of surgery
  Operator experience will be assessed as the number of years of clinical experience performing periodontal or soft tissue grafting procedures. Higher numbers indicate greater operator experience.
  Unit of Measure: Years of clinical experience
Healing of the donor site | 1-week and 2-weeks post-surgery
  Healing of the donor site will be assessed using a modified wound healing score with four variables: Necrosis, Fibrin/Granulation Tissue, Bleeding on Palpation, and Texture, each scored 0-2:
  Variable: 0 1 2 Necrosis: Complete Incomplete Absent Fibrin/Granulation Tissue: Fibrin > granulation tissue Fibrin = granulation tissue Fibrin < granulation tissue Bleeding on Palpation: Present Slight Absent Texture: Obvious difference Moderate difference No difference
  Two blinded clinical examiners will independently evaluate standardized photographs at 1 week and 2 weeks postoperatively. Higher total scores indicate better wound healing. Inter-rater reliability will be calculated.
  Unit of Measure: Score (0-8), sum of four variables on the modified wound healing score

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universitària d'Odontologia - UIC Barcelona, Barcelona, Sant Cugat Del Valles, Spain

IPD SHARING:
Plan to Share IPD: No